CLINICAL TRIAL: NCT01910792
Title: Ultraviolet Light and Vitamin D in Subjects With Fat Malabsorption or After Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Michael F. Holick, PhD, MD, Boston University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-30047
Record Dates: First submitted 2012-06-25; First posted 2013-07-30 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Vitamin D Deficiency; Gastrointestinal Diseases
MeSH Terms: conditions — Vitamin D Deficiency; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 2 (Active Comparator): Patients who have had gastric bypass surgery will be exposed to a Sperti Lamp 3x/week
  Interventions: Device: Sperti Lamp
- Group 1 (Active Comparator): Patients with fat malabsorption syndromes will be exposed to a Sperti Lamp 3x/week
  Interventions: Device: Sperti Lamp

INTERVENTIONS:
Device: Sperti Lamp — UV light exposure 3 times per week for 12 weeks

SUMMARY:
Patients with fat malabsorption due to Crohn's disease, ulcerative colitis, or other causes including cystic fibrosis, among others, or who have undergone gastric bypass have increased incidence of vitamin D deficiency relative to the general population. Given that vitamin D is fat soluble and absorbed in the proximal small intestine, it has been documented that vitamin D deficiency in people with a fat malabsorption syndrome is due to decreased absorption of vitamin D.

The amount of vitamin D produced from winter sunlight (in Boston, MA) and dietary sources will negligibly raise blood vitamin D levels in these patients, and oral vitamin D supplementation may have limited efficacy due to malabsorption. A variety of UV light sources have been developed and sold as in-home tanning devices and to produce vitamin D in reptiles. The efficacy of correcting vitamin D deficiency by the skin exposure to an artificial source of UVB radiation in patients with fat malabsorption syndromes (Crohn's disease, ulcerative colitis, or cystic fibrosis) or after gastric bypass surgery has not been studied. The investigators have conducted a pilot study in healthy adults that demonstrated that exposure to the lamp raised the blood level of 25-hydroxyvitamin D with no side effects. The main purpose of this study is to evaluate the effect of the FDA approved artificial source of ultraviolet (UVB) radiation (Sperti® lamp) in improving vitamin D status in patients with fat malabsorption syndromes and patients who have undergone roux-en-Y gastric bypass surgery.

DETAILED DESCRIPTION:
Given that vitamin D is absorbed in the proximal small intestine, it is believed that vitamin D deficiency in people with a fat malabsorption syndrome may be due to decreased absorption of vitamin D. All diseases of the small bowel can cause fat malabsorption. These fat malabsorption syndromes include Crohn's disease, ulcerative colitis, or cystic fibrosis among others (1,2) and affect the amount of nutrients and fat absorbed by the gastrointestinal tract.

Gastric bypass surgery is indicated for the surgical treatment of morbid obesity by making the stomach smaller and allowing food to bypass proximal part of the small intestine, where many minerals and vitamins are most absorbed. Food (and calorie) intake is dramatically reduced because of the new small stomach. Many patients who have bypass surgery develop nutritional deficiencies because they do not adhere to their post-operative guidelines concerning the need for nutritional supplements. Malabsorptive operations like gastric bypass surgery pose a particular risk for multiple nutritional deficiencies, including vitamin D malabsorption. (3) Vitamin D is ingested in the diet, from supplements, as well as synthesized naturally in the skin following UVB irradiation from the sun. As sunlight enters the atmosphere, all radiation below 290 nm is absorbed by the stratospheric ozone layer. Radiation between 290 and 315 nm is responsible for converting 7-dihydrocholesterol (provitamin D3) in the epidermis and dermis to previtamin D3. Once formed, previtamin D3 undergoes a thermally induced isomerization to vitamin D3. Vitamin D3 enters the circulation and is metabolized in the liver to 25-hydroxyvitamin D3 [25(OH)D] and then in the kidney to 1,25-dihydroxyvitamin D3 [1,25(OH)2D] by the 25-hydroxyvitamin D3-1á-hydroxylase [1á-OHase]. 25(OH)D is the major circulating form of vitamin D and is routinely measured in the blood to determine the vitamin D status of a patient.

The amount of vitamin D produced from winter sunlight and dietary sources will negligibly raise blood 25-hydroxy vitamin D levels. People living in areas that receive less sunlight have lower circulating 25-hydroxyD (the major circulating form used to measure vitamin D status) levels. Vitamin D deficiency (defined as a serum 25(OH)D level < 20 ng/ml) in the general population is treated with oral supplementation of vitamin D at a dose of 50,000 IU given once weekly for eight weeks. (1) However from clinical experiences, oral supplementation has limited efficacy in vitamin D deficiency patients with malabsorption syndromes likely due to the inability to efficiently absorb vitamin D. *(1-3) A variety of UV light sources have been developed and sold as in-home tanning devices and to produce vitamin D in reptiles. In a pilot study, the investigators have observed that 5 out of 8 subjects had significant increased circulating 25(OH)D after exposure to a Sperti® lamp for 24 weeks. However, the possibility of correcting vitamin D deficiency by the skin exposure to artificial source of UVB radiation in patients with fat malabsorption has not been studied.

The first aim of this study will be to evaluate the efficacy of an FDA approved artificial source of UVB radiation (Sperti® lamp) in raising serum 25(OH)D levels in patients with fat malabsorption due to Crohn's disease, ulcerative colitis, or cystic fibrosis or gastric bypass surgery and other causes. The second aim of the study is to compare the rise in serum 25(OH)D over the repeated measures in this study in patients with the 4 different skin types (types II-V).

The device that the investigators used in this study was originally designed for tanning. From our pilot study H23521 the investigators observed that much longer times were needed to increase the production of vitamin D. As can be seen in Figure 1, our healthy adults exposed to up to 10 minutes to the Sperti lamp showed significant increases in serum 25 (OH)D levels in the subjects studied. The investigators found that 5 of the 8 subjects showed significant increases in 25(OH)D. Those with skin type IV and V demonstrated minimal responses due to the sunscreening effect of their skin pigment (Fig 2). This demonstrates that skin types IV and V may require longer exposure times to achieve the 0.75 MED dose and raise the serum 25(OH)D level. However, during this pilot study, the investigators did not observe any untoward side effects (such as skin redness) associated with exposure to UVB light with longer exposure times.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 18 years or older with skin types 2,3,4 and 5.
2. The patient has an established diagnosis of conditions that have been associated with fat malabsorption due to bowel disease (Crohn's disease, ulcerative colitis, or cystic fibrosis), or history of gastric bypass surgery that at least 3 months post-surgery with no continuing complications.
3. The patient is able to understand the information provided to them and who have given written informed consent to the study.
4. The patient is able to understand and complete self-administered questionnaires.
5. The patient is able and willing to follow study procedures.
6. If female, the patient is either postmenopausal for at least one year, surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (oral or parenteral hormonal contraceptive; intrauterine device; barrier and spermicide or abstinence). Patients must agree to use adequate contraception during the study.

Exclusion Criteria:

1. Treatment with pharmacologic doses of vitamin D3, vitamin D3 metabolites or analogues, ongoing or within 30 days prior the start of the study.
2. Pregnancy and lactation.
3. History of underlying photosensitivity.
4. Patients with a history of chronic kidney disease or severe liver dysfunction that would alter their calcium and vitamin D metabolism.
5. Subjects with skin type I (who will develop skin burns after UVB exposure).
6. Use of medications that cause a photosensitivity reaction including hydrochlorothiazide or tetracycline.
7. History of skin cancer .
8. Patients with history of hypocalcemia (calcium <8.6mg%), hypercalcemia (calcium >10.4mg%).
9. Taking drugs known to influence vitamin D metabolism, such as glucocorticoids and antiseizure medications.
10. Patients with a history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease within 3 months.
11. Patients who have travelled through a warm sunny climate without using sunscreen within 1 month of the beginning of the study, or plan to do so during the study period.
12. Patients who taking any medications which causes skin sensitivity to sunlight (certain antibiotics; retin-A cream used for acne).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Holick, PhD, MD, Principal Investigator — BUMC
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be recruited from the Center for Digestive Disorders or the Endocrinology, Diabetes, and Nutrition clinic during regularly scheduled outpatient visits. Subjects will also be recruited by placing IRB approved posters around BUMC and also placing an IRB approved email in the monthly resear
Groups:
- Pts w/ Gastric Bypass: Patients who have had gastric bypass surgery will be exposed to a Sperti Lamp 3x/week
  Sperti Lamp: UV light exposure 3 times per week for 12 weeks
- Pts w/ Fat Malabsorption: Patients with fat malabsorption syndromes will be exposed to a Sperti Lamp 3x/week
  Sperti Lamp: UV light exposure 3 times per week for 12 weeks
Period: Overall Study
Arm/Group | Pts w/ Gastric Bypass | Pts w/ Fat Malabsorption
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 2 | Group 1 | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
Established diagnosis of Fat Malabsorption Syndromes [Count of Participants; unit: Participants] | 0 | 10 | 10
History of Gastric Bypass at least 3 months post-op with no continuing complications [Count of Participants; unit: Participants] | 9 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: # of Pts w/ Enhanced Vitamin D Status
Description: Increase circulating 25(OH)D levels
Time Frame: Baseline, Months 1, 2, 3
Population: Only 3 subjects in each Arm had a conclusive set of data eligible for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pts w/ Gastric Bypass | Pts w/ Fat Malabsorption
Number analyzed (Participants) | 3 | 3
Participants | 3 | 3

ADVERSE EVENTS:
Arm/Group | Pts w/ Gastric Bypass | Pts w/ Fat Malabsorption
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No